CLINICAL TRIAL: NCT00757952
Title: Early Detection of Epithelial Ovarian Cancer Using Exhaled Breath Markers: GC/FT-ICR Mass Spectrometry and Canine Olfaction.
Brief Title: Early Detection of Ovarian Cancer: GC/FT-ICR Mass Spectrometry and Canine Olfaction
Status: Completed | Type: Observational
Sponsor: Pine Street Foundation (Other)
Responsible Party: Principal Investigator, Michael McCulloch, Principal Investigator, Pine Street Foundation
Other Study IDs: PINE-A-14183; CDR0000614811 (Registry Identifier: PDQ (Physician Data Query)); UCSF-H105-31440-01
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Chromatography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fourier transform ion cyclotron resonance mass spectrometry
Other: chromatography
Other: diagnostic laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of exhaled breath from patients with ovarian epithelial cancer, polycystic ovarian syndrome, or endometriosis and from healthy participants in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors find and diagnose ovarian epithelial cancer sooner, when it may be easier to treat.

PURPOSE: This clinical trial is studying exhaled breath biomarkers to see how well they find ovarian epithelial cancer in patients with newly diagnosed ovarian epithelial cancer, polycystic ovarian syndrome, or endometriosis and in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify patterns of exhaled compounds in breath samples from patients with newly diagnosed ovarian epithelial cancer that are significantly and reproducibility different from those of healthy volunteers using gas chromatography Fourier transform ion cyclotron resonance mass spectrometry (GC/FT-ICR MS).
* Train five canines to discriminate between exhaled breath samples from patients with newly diagnosed ovarian epithelial cancer and healthy volunteers.
* Use both canine olfaction and GC/FT-ICR MS to distinguish between exhaled breath samples from patients with newly diagnosed ovarian epithelial cancer and patients with polycystic ovarian syndrome or endometriosis.
* Repeat breath sampling in patients with newly diagnosed ovarian epithelial cancer throughout the course of diagnosis and therapy.

OUTLINE: Exhaled breath samples are collected from patients and healthy volunteers. The samples are analyzed by gas chromatography Fourier transform ion cyclotron resonance mass spectrometry (GC/FT-ICR MS) to determine chemical compositions, identities, and predictive patterns of biomarkers in exhaled breath condensate. GC/FT-ICR MS and trained canine olfaction are used to distinguish between exhaled breath samples from patients with ovarian epithelial cancer, patients with polycystic ovarian syndrome or endometriosis, and healthy volunteers.

Patients and healthy volunteers complete questionnaires about BRCA 1 and BRCA 2 status (if known), alcohol use, smoking (including duration and type of cigarettes), physical activity (duration and type), socioeconomic status, education, county of residence, age at menopause (if applicable), age at menarche, presence of first- and second-degree family history of breast cancer or ovarian epithelial cancer, body mass index (height and weight), and co-morbidities.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets one of the following criteria:

  * Histologically confirmed ovarian epithelial cancer

    * Newly diagnosed disease
  * Diagnosis of polycystic ovarian syndrome or endometriosis
  * Healthy volunteer meeting all of the following criteria:

    * No prior ovarian cancer (including invasive ovarian epithelial cancer, fallopian tube cancer, or primary papillary serous carcinoma of the peritoneum)
    * No prior breast cancer (including ductal carcinoma in situ [DCIS])
    * No prior ovarian or breast cancer (including DCIS) in any first- or second-degree relative
    * BRCA1 or BRCA2 mutation negative (if known) OR no first- or second-degree relative with a BRCA1 or BRCA2 mutation (if known)
* No prior diagnosis of cancer

PATIENT CHARACTERISTICS:

* Lives in California and close to the study sampling centers
* Reads and writes English, Spanish, or Chinese
* Non-smoker
* Willing to provide breath samples
* No alcohol intake within the past 3 days

PRIOR CONCURRENT THERAPY:

* At least 3 days since prior Cox-2 inhibitors, vitamin E, omega-3 fatty acids, antioxidants, bromelain, coenzyme Q10, curcumin, or vitamin A

Ages: 21 Years to 120 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Histologically confirmed ovarian epithelial cancer.
  2. Polycystic Ovarian Syndrome or Endometriosis
  3. Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2007-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Identification of patterns of exhaled compounds in breath samples using gas chromatography Fourier transform ion cyclotron resonance mass spectrometry (GC/FT-ICR MS) | 2009-2012
Diagnostic accuracy of GC/FT-ICR MS in distinguishing between exhaled breath samples from patients with ovarian epithelial cancer, patients with polycystic ovarian syndrome or endometriosis, and healthy volunteers | 2009-2012
Diagnostic accuracy of canine scent detection in distinguishing between exhaled breath samples from patients with ovarian epithelial cancer and healthy volunteers | 2009-2012

CONTACTS AND LOCATIONS:
Overall Officials: Michael McCulloch, MPH, PhD, Principal Investigator — Pine Street Foundation
Locations (4):
- United States (4):
  - Pine Street Foundation, San Anselmo, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - University of Maine, Orono, Maine